CLINICAL TRIAL: NCT02726958
Title: Early Postoperative Blood Glucose Variability and Outcome After TAVI : a Retrospective Single-centre Study
Brief Title: Early Postoperative Blood Glucose Variability and Outcome After TAVI
Acronym: GLYTAVI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Guillaume BESCH, M.D., Centre Hospitalier Universitaire de Besancon
Other Study IDs: EI/2014/141
Record Dates: First submitted 2016-03-30; First posted 2016-04-04 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Stress Hyperglycemia
Keywords: aortic valve replacement; percutaneous valve; blood glucose variability; TAVI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- group M: patients who died or suffered from stroke, acute coronary syndrome, heart failure, complete atrioventricular block or life-threatening ventricular arrhythmias within 30 days after the procedure
- group T: other patients

SUMMARY:
Stress hyperglycaemia is a well-known risk factor of postoperative morbidity and mortality in cardiac surgery. Recently, several authors have reported that increased blood glucose (BG) variability could worsen the prognosis in this population.The transcatheter aortic valve implantation (TAVI) is a low invasive procedure proposed as an alternative technique to aortic valve replacement surgery in high-risk patients.

The aim of this study is to describe the incidence of stress hyperglycaemia and assess whether BG variability could impact the outcome of patients undergoing TAVI.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years old
* severe degenerative symptomatic aortic stenosis
* logistic Euroscore ≥ 20% or/and Society of Thoracic Surgeons score (STS) ≥ 10%
* recused for a conventional valve replacement by multidisciplinary team (surgeon, cardiologist) because of surgical contraindication or comorbidities related to the patient.
* written consent before the procedure concerning anonymous data processing.

Exclusion Criteria:

* death per procedure
* postoperative admission in a critical care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Planned transcatheter aortic valve implantation
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Incidence of stress hyperglycemia | 48 hours
  Stress hyperglycemia is defined as a blood glucose value above 7.7 mmol/l requiring insulin infusion within the 48 first hours following the TAVI.

SECONDARY OUTCOMES:
Mean blood glucose value | 48 hours
  Mean blood glucose value is the mean of all the blood glucose values measured during the 48 first hours following the TAVI.
Standard deviation of blood glucose value | 48 hours
  Standard deviation of glucose value is the standard deviation of all the blood glucose values measured during the 48 first hours following the TAVI.
Incidence of moderate hypoglycemia | 48 hours
  Moderate hypoglycemia is defined as a blood glucose value under 3.3 mmol/l.
Incidence of severe hypoglycemia | 48 hours
  Severe hypoglycemia is defined as a blood glucose value under 2.2 mmol/l.
Incidence of severe hyperglycemia | 48 hours
  Severe hyperglycemia is defined as a blood glucose value above 11.0 mmol/l.
Coefficient of variability of blood glucose | 48 hours
  The coefficient of variability is the ratio of the standard deviation on the mean blood glucose value, expressed as a percentage.
Mean daily variation of blood glucose | 48 hours
  The mean daily variation of blood glucose is defined as the mean of the daily differences between the maximal and the minimal glucose value.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie DEPIERRE, Study Chair — Centre hospitalier régional universitaire de Besançon
Locations (1):
- CHRU Jean Minjoz Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldberg PA, Sakharova OV, Barrett PW, Falko LN, Roussel MG, Bak L, Blake-Holmes D, Marieb NJ, Inzucchi SE. Improving glycemic control in the cardiothoracic intensive care unit: clinical experience in two hospital settings. J Cardiothorac Vasc Anesth. 2004 Dec;18(6):690-7. doi: 10.1053/j.jvca.2004.08.003. PMID 15650975
- [Background] Meyfroidt G, Keenan DM, Wang X, Wouters PJ, Veldhuis JD, Van den Berghe G. Dynamic characteristics of blood glucose time series during the course of critical illness: effects of intensive insulin therapy and relative association with mortality. Crit Care Med. 2010 Apr;38(4):1021-9. doi: 10.1097/CCM.0b013e3181cf710e. PMID 20124887
- [Background] Dossett LA, Cao H, Mowery NT, Dortch MJ, Morris JM Jr, May AK. Blood glucose variability is associated with mortality in the surgical intensive care unit. Am Surg. 2008 Aug;74(8):679-85; discussion 685. doi: 10.1177/000313480807400802. PMID 18705566
- [Background] Bagshaw SM, Bellomo R, Jacka MJ, Egi M, Hart GK, George C; ANZICS CORE Management Committee. The impact of early hypoglycemia and blood glucose variability on outcome in critical illness. Crit Care. 2009;13(3):R91. doi: 10.1186/cc7921. Epub 2009 Jun 17. PMID 19534781
- [Background] Egi M, Bellomo R, Reade MC. Is reducing variability of blood glucose the real but hidden target of intensive insulin therapy? Crit Care. 2009;13(2):302. doi: 10.1186/cc7755. Epub 2009 Apr 6. PMID 19435472
- [Background] Gilard M, Eltchaninoff H, Iung B, Donzeau-Gouge P, Chevreul K, Fajadet J, Leprince P, Leguerrier A, Lievre M, Prat A, Teiger E, Lefevre T, Himbert D, Tchetche D, Carrie D, Albat B, Cribier A, Rioufol G, Sudre A, Blanchard D, Collet F, Dos Santos P, Meneveau N, Tirouvanziam A, Caussin C, Guyon P, Boschat J, Le Breton H, Collart F, Houel R, Delpine S, Souteyrand G, Favereau X, Ohlmann P, Doisy V, Grollier G, Gommeaux A, Claudel JP, Bourlon F, Bertrand B, Van Belle E, Laskar M; FRANCE 2 Investigators. Registry of transcatheter aortic-valve implantation in high-risk patients. N Engl J Med. 2012 May 3;366(18):1705-15. doi: 10.1056/NEJMoa1114705. PMID 22551129
- [Background] Eltchaninoff H, Prat A, Gilard M, Leguerrier A, Blanchard D, Fournial G, Iung B, Donzeau-Gouge P, Tribouilloy C, Debrux JL, Pavie A, Gueret P; FRANCE Registry Investigators. Transcatheter aortic valve implantation: early results of the FRANCE (FRench Aortic National CoreValve and Edwards) registry. Eur Heart J. 2011 Jan;32(2):191-7. doi: 10.1093/eurheartj/ehq261. Epub 2010 Sep 15. PMID 20843959
- [Derived] Besch G, Pili-Floury S, Morel C, Gilard M, Flicoteaux G, Salomon du Mont L, Perrotti A, Meneveau N, Chocron S, Schiele F, Le Breton H, Samain E, Chopard R. Impact of post-procedural glycemic variability on cardiovascular morbidity and mortality after transcatheter aortic valve implantation: a post hoc cohort analysis. Cardiovasc Diabetol. 2019 Mar 11;18(1):27. doi: 10.1186/s12933-019-0831-3. PMID 30857532